CLINICAL TRIAL: NCT02008149
Title: Using Musculoskeletal Models to Assess FES Rowing for Skeletal Health After SCI
Brief Title: FES Rowing for Skeletal Health After SCI
Acronym: FES-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1410-P; 5I21RX001410-02 (NIH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injury
Keywords: Osteoporosis
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Group assignment will be based on the preference of potential subjects. Subjects can either participate in the FES-rowing group or they can participate in the standard-of-care group. The standard-of-care group will not perform FES-rowing; they will only receive periodic bone density measurements over a 36-week period, with a total time commitment of approximately 10 hours. Subjects in the FES-rowing group will participate in rowing sessions requiring a 2 to 3 hour time commitment per week for the duration of the participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care group (No Intervention): SCI individuals receiving conventional rehab
- FES-rowing group (Experimental): Individuals with SCI participating in an FES-rowing program
  Interventions: Other: Rowing exercise

INTERVENTIONS:
Other: Rowing exercise — Individuals with SCI will use the rowing exerciser to see if there is a benefit to skeletal health in the lower limbs.
  Arms: FES-rowing group

SUMMARY:
Following a complete spinal cord injury (SCI), individuals experience progressive bone loss, especially in the legs, with up to 70% of persons with SCI sustaining a fracture at some point during their lifetime. Fractures following SCI are costly to treat and more than half of patients experience a medical complication, requiring extended hospitalization, resulting in a substantial impact on their quality of life. To reduce the incidence of fractures, more effective rehabilitation strategies to prevent bone loss are needed. The goal of this research is to determine if bone health can be preserved using an indoor rowing exercise program in which the leg muscles are electrically stimulated using several, small surface electrode pads that are placed on the skin on the front and back thigh muscles. An encouraging case study has recently shown remarkable bone preservation in one individual with SCI who participated in an electrical stimulation rowing program, however, whether other individuals with SCI can achieve the same benefit is currently unknown.

DETAILED DESCRIPTION:
In this study the investigators expect to enroll a total of 10 participants with SCI. Five participants will be assigned to a Standard-of-Care (control) group and five participants will be assigned to an FES-rowing intervention group. Group assignment will be partly based on the preference of each potential participant and their willingness to make the necessary time commitment required for participation in a given group, with the added goal, to the extent possible, of matching the two groups for age, gender and time since injury. Only those individuals who have a strong desire to participate in a regular exercise program and who express a willingness to travel to VA Palo Alto the necessary number of times per week to perform FES-rowing will be potential candidates for inclusion in the rowing group.

Bone density measurements for both the Standard-of-Care group and the FES-rowing group will be performed using Dual energy X-ray Absorptiometry (DXA) and peripheral Quantitative Computed Tomography (pQCT). The Standard-of-Care group will undergo no other research procedures.

The muscle conditioning program is accomplished through electrical stimulation of the quadriceps and hamstring muscles using a 4-channel electrical stimulator that applies stimulation using surface electrodes adhered using gel to the skin overlying the quadriceps and hamstrings muscles. The muscle strengthening initially takes place three times per week, sixty minutes per session, progressing up to five sessions per week, for approximately 8 weeks. The muscle strengthening program ensures that subjects have sufficient muscle strength and endurance before they embark on the rowing program. Following the 8-week muscle strengthening program, subjects will begin FES-rowing, with three sessions per week, thirty minutes per session for the following 28 weeks. In the FES-rowing group, the investigators will measure isometric knee extension strength at the start of week 0, and at the end of weeks 12, 24 and 36.

For the rowing group, the investigators will capture 3D kinetics and kinematics in the motion capture laboratory during FES-rowing at the end of weeks 12, 24 and 36. Kinematics during rowing will be collected from fifty passive retro-reflective markers that will be placed on each participant to capture the position and orientation of the 12 interconnected body segments used to represent each subject.

ELIGIBILITY:
Inclusion Criteria:

Subjects in the rowing groups:

* male and female SCI outpatients or inpatients
* have a C7 to T12, ASIA-A or ASIA-B, spinal cord injury
* be at least 18 years old
* have their physician's clearance to exercise
* between 3 and 24 months post spinal cord injury*
* minimum passive hip flexion range of motion (ROM) from 20 to 100 deg
* minimum passive knee flexion ROM from 20 to 100 deg
* minimum passive ankle ROM from +10 deg (dorsi-flexion) to -15 deg (plantar-flexion)
* currently use a manual wheelchair
* be able to perform independent and safe transfers to and from their wheelchair *There is no time post injury restriction for subjects in the experience rower group

Subjects in the control group:

* male and female SCI outpatients or inpatients
* have a C5 to T12, ASIA-A or ASIA-B, spinal cord injury
* be at least 18 years old
* between 3 and 24 months post spinal cord injury
* be able to perform safe transfers to and from their wheelchair, either independently or with assistance

Exclusion Criteria:

* pregnant women
* women of childbearing potential not practicing a reliable method of contraception
* women who are post-menopausal
* have mechanical instability of the spine
* resting blood pressure higher than 140/90
* a grade 1 or greater, sacral, gluteal or ischial pressure ulcer
* history of low trauma, lower limb fracture since SCI
* renal disease
* current osteomyelitis
* current thrombosis/hemorrhage
* cancer
* other neurological disease (i.e. stroke, peripheral neuropathy, myopathy)
* any implanted electronic device
* active treatment for epilepsy
* regular use of tobacco
* known coronary artery disease
* family history of sudden cardiac death
* current use of cardioactive medications, e.g., for treatment of congestive heart failure or arrhythmia
* current use of medications that can affect bone density and fracture risk including:

  * bisphosphonates
  * parathyroid hormone (PTH) and PTH analogs
  * androgenic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Beaupre, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lambach RL, Stafford NE, Kolesar JA, Kiratli BJ, Creasey GH, Gibbons RS, Andrews BJ, Beaupre GS. Bone changes in the lower limbs from participation in an FES rowing exercise program implemented within two years after traumatic spinal cord injury. J Spinal Cord Med. 2020 May;43(3):306-314. doi: 10.1080/10790268.2018.1544879. Epub 2018 Nov 26. PMID 30475172

RESULTS

PARTICIPANT FLOW:
Groups:
- FES-Rowers: Individuals with complete SCI participating in a 90-session FES-rowing program.
- Standard-of-Care Controls: Individuals with complete SCI undergoing bone density scanning at four time points over 9 months.
- Experienced FES-Rower: An individual with more than 10 years of FES-Rowing experience.
Period: Overall Study
Arm/Group | FES-Rowers | Standard-of-Care Controls | Experienced FES-Rower
Started | 7 | 1 | 1
Completed | 4 | 0 | 1
Not Completed | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FES-Rowers | Standard-of-Care Controls | Experienced FES-Rower | Total
Number analyzed (Participants) | 7 | 1 | 1 | 9
Age, Continuous [Mean (Full Range); unit: Years] | 33 [23 to 43] | 24 [24 to 24] | 59 [59 to 59] | 35 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 1 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 1 | 0 | 8
  United Kingdom | 0 | 0 | 1 | 1
Baseline Bone Mineral Density [Mean (Full Range); unit: g/cm^3] — 4% distal femur bone mineral density (g/cm^3) from peripheral quantitative computed tomography scanning
  g/cm^3 | 216.1 [142.9 to 262.0] | 227.3 [227.3 to 227.3] | 251.2 [251.2 to 251.2] | 221.3 [142.9 to 262.0]

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: Bone mineral density at the distal femur at 0, 16, 29 and 43 weeks measured using peripheral quantitative computed tomography scanning.
Time Frame: 0, 16, 29 and 43 weeks
Population: The only participant in the Stanford-of-Care Control group self-withdrew after 12 weeks of participation, after having a baseline measurement and one other bone density measurement. The participant in the Experienced FES-Rower group was only measured at baseline.
Measure: Mean (Full Range); unit: g/cm^3
Arm/Group | FES-Rowers | Standard-of-Care Controls | Experienced FES-Rower
Number analyzed (Participants) | 7 | 1 | 1
g/cm^3
  Bone Mineral Density at 16 wks: number analyzed (Participants) | 6 | 0 | 0
  Bone Mineral Density at 16 wks | 184.0 [127.8 to 238.5] |  |
  Bone Mineral Density at 29 wks: number analyzed (Participants) | 5 | 0 | 0
  Bone Mineral Density at 29 wks | 174.9 [97.2 to 229.6] |  |
  Bone Mineral Density at 43 wks: number analyzed (Participants) | 4 | 0 | 0
  Bone Mineral Density at 43 wks | 188.5 [141.8 to 229.5] |  |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | FES-Rowers | Standard-of-Care Controls | Experienced FES-Rower
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/7 | 0/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FES-Rowers (N=7) | Standard-of-Care Controls (N=1) | Experienced FES-Rower (N=1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Muscle strain from hand cycling unrelated to study

LIMITATIONS AND CAVEATS:
Small number of FES-rowers was due to the time commitment of approximately 138 hours over a 9-12 month period..

Small number of subjects in the Standard-of-Care group was due to the 9-12 month time commitment and the lack of perceived benefits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT02008149/Prot_SAP_ICF_000.pdf